CLINICAL TRIAL: NCT06646692
Title: Mindful Self-Compassion to Address PTSD and Substance Use in Unhoused Women
Acronym: MSC for PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Dana Rose Garfin, Associate Professor-in-Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-000260; W911NF-23-1-0208:P00002 (Other Grant/Funding Number: DOD-DA-U.S. Army Contracting Command (USACC))
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Posttraumatic Stress Disorder (PTSD); Anxiety; Depression - Major Depressive Disorder
Keywords: homelessness; mindful self compassion; depression; substance use disorder; craving; PTSD; posttraumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression; Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Self Compassion Classes (Experimental): (MSC) is a mind-body integrative health intervention that utilizes meditations, other contemplative practices, home practices, and experiential exercises (including group discussions) to increase SC. MSC can be done in groups of 10-25. To increase feasibility of MSC for use in residential drug treatment facilities we will aim to adapt MSC to 7 sessions (6 weekly sessions in alignment with the MSC short course plus the half day retreat included in the full course to facilitate skill consolidation). Sessions will be conducted in a group-based format: prior research found group-based formats equivalent to individual-level interventions for PTSD/SUD.
  Interventions: Behavioral: Mindful Self Compassion
- Treatment as Usual (Experimental): Selecting appropriate attention control groups for behavioral intervention research, particularly for mindfulness-based interventions, can be problematic. Comparator groups often also improve as they tend to target related mechanisms (e.g., social support, health behaviors, improved attention). After weighing the pros and cons, a "treatment as usual" (TAU) approach was selected, whereby the MSC will be compared to TAU. However, to control for the confound of weekly compensation, TAU participants will meet with study staff seven times over the 6-week period and fill out short psychosocial surveys on non-distressing topics (e.g., personality tests, attitudes surveys) in exchange for compensation commensurate with the MSC group. We believe this will also help with retention of the TAU group over time and strike an appropriate balance between controlling for the effects of study participation while minimizing confounds that often occur with active control groups in behavioral trials.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Mindful Self Compassion — (MSC) is a mind-body integrative health intervention that utilizes meditations, other contemplative practices, home practices, and experiential exercises (including group discussions) to increase SC. MSC can be done in groups of 10-25. To increase feasibility of MSC for use in residential drug treatment facilities, we will aim to adapt MSC to 7 sessions (6 weekly sessions in alignment with the MSC short course plus the half day retreat included in the full course to facilitate skill consolidation). Sessions will be conducted in a group-based format: prior research found group-based formats equivalent to individual-level interventions for PTSD/SUD.
  Other Names: MSC
  Arms: Mindful Self Compassion Classes
Behavioral: Treatment as Usual (TAU) — Selecting appropriate attention control groups for behavioral intervention research, particularly for mindfulness-based interventions, can be problematic. Comparator groups often also improve as they tend to target related mechanisms (e.g., social support, health behaviors, improved attention). After weighing the pros and cons, a "treatment as usual" (TAU) approach was selected, whereby the MSC will be compared to TAU. However, to control for the confound of weekly compensation, TAU participants will meet with study staff seven times over the 6-week period and fill out short psychosocial surveys on non-distressing topics (e.g., personality tests, attitudes surveys) in exchange for compensation commensurate with the MSC group. We believe this will also help with retention of the TAU group over time and strike an appropriate balance between controlling for the effects of study participation while minimizing confounds that often occur with active control groups in behavioral trials.
  Other Names: TAU
  Arms: Treatment as Usual

SUMMARY:
Trauma exposure, posttraumatic stress disorder (PTSD), and substance use disorder (SUD) present major threats to public health. PTSD and SUD are major correlates of disability, often resulting in severe social and occupational impairment. Comorbidity between PTSD and SUD (PTSD/SUD) is common and frequently co-occurs with other mental health ailments including depression, anxiety, and suicidality. Comorbidity may be amplified in groups vulnerable to high trauma exposure, such as women with low socioeconomic status including women experiencing homelessness (WEH). Moreover, the reciprocal nature of PTSD/SUD (substances are used to cope with PTSD symptoms; substance use can create high-risk situations for new traumas to occur), can create a cycle of trauma and symptomatology leading to a critical health disparity.

PTSD/SUD can be costly and difficult to treat, with treatment completion often low and relapse rates often high. Low-cost, complementary interventions, such as self-compassion (SC) interventions, which target key mechanisms that maintain PTSD/SUD, could improve treatment outcomes. SC interventions include practices that build skills to improve emotional responses, cognitive understanding, and mindfulness. Recent research supports the benefit of SC interventions for reducing PTSD, SUD, and related comorbidities, potentially with large effects. However, sample sizes have generally been small and randomized designs infrequently used. Moreover, while SC interventions may act to improve key mechanisms of treatment response and/or symptom maintenance (e.g., emotion regulation/dysregulation, trauma-related guilt, trauma-related shame, moral injury, and craving), such mediating factors have been underexplored. To address these limitations, the present proposal will implement community-based research principles and use a two phase, mixed-method design to adapt and test a widely used SC intervention (Mindful Self Compassion; MSC) for use with a sample of WEH with PTSD/SUD. The project will be conducted in partnership with a state-funded drug treatment facility that serves women and families experiencing high health disparities.

Phase I was completed in 2023 and adapted the standard MSC course for use with trauma-exposed WEH with PTSD/SUD using the ADAPT-ITT model, an eight-stage model that engages community partners to increase feasibility and acceptability of interventions for at-risk populations.

Phase II will be an open-label cluster randomized clinical trial (N=202) to test the benefit of the adapted MSC at improving primary (PTSD, substance use) and secondary outcomes (depression, anxiety, hopelessness) among a sample of WEH with PTSD/SUD residing in a residential drug treatment site. MSC (n=101) will be compared to Treatment as Usual (TAU; n=101). WEH in the MSC group will complete a 6-week (six sessions plus a half-day retreat) MSC intervention.

The TAU group will engage in weekly check-ins with the research team but will not receive an intervention. WEH will be assessed at baseline, immediately post-intervention, and at a 4-month follow-up. One-on-one interviews will be conducted with the MSC group to collect qualitative data on experiences. An exploratory aim will be to elucidate mechanism of treatment-response and maintenance or remission of PTSD symptoms. These potential mechanisms will include SC, emotion regulation/dysregulation, trauma-related guilt, trauma-related shame, moral injury, and craving.

Results may inform treatment for PTSD/SUD in WEH and other groups experiencing high health disparities and provide valuable insights into mechanisms underlying PTSD/SUD symptoms over time. Findings are relevant to military populations, which experience high rates of PTSD/SUD, and other populations disproportionately exposed to trauma.

ELIGIBILITY:
Inclusion Criteria:

* Identifies as woman
* Age 18 and over
* Probable PTSD as judged by the PCL-5 (score of 31 or higher, indicated as having optimal signal detection)
* No cognitive impairment according to a score of < 10 on the Short-Blessed Test
* Experienced homelessness in the past 6 months or prior to incarceration ("spent night in public or private shelter or on the street")
* Able to speak and understand English.

Exclusion Criteria:

* Not able to speak English
* Judged to be cognitively impaired, as indicated by score > 10 on the Short-Blessed Screener
* Does not meet other inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological women or individuals who identify as a woman are eligible to participate in the study
Enrollment: 202 (Estimated)
Dates: Start 2024-05-05 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
PTSD | T1 (baseline, enrollment), T2 (immediate follow-up), T3 (4-months post-baseline)
  PTSD symptoms will be measured using the PTSD Checklist for Diagnostic and Statistical Manuel of Mental Disorders, DSM-5 (PCL-5), which will be scored continuously and according to diagnostic criteria.2 The PCL-5 initially starts with the identification of the presence of exposure to a Diagnostic and Statistical Manual of Mental Disorders, DSM-V traumatic event; assesses actual or threatened death, serious injury or sexual violence; and whether the person directly experienced it. Twenty additional items assess all four B-E criteria (re-experiencing, avoidance, negative thoughts or cognitions, hyperarousal), assessed on a Likert-type scale from 0 (not at all) to 4 (extremely). Treatment response will be defined as a ≥ 5-point reduction in symptoms and clinically meaningful improvement as ≥ 10-point reduction in symptoms. PTSD will be assessed for worse lifetime event and (if applicable) worst event in the past year.
Alcohol Use Disorders Identification Test (AUDIT) | T1 (baseline, enrollment), T2 (immediate follow-up), T3 (4-months post-baseline)
  The AUDIT is part of the National Institute on Drug Abuse (NIDA) Clinical Trials Network (CTN) Common Data Elements for use in clinical trials. The Audit is a 10-item alcohol screen that helps identify persons who are hazardous drinkers or who have active alcohol use disorders. It can be calculated as a sum score and will be analyzed as a continuous and categorical (yes/no used alcohol) outcome.
Drug Abuse Screening Test (DAST) | T1 (baseline, enrollment), T2 (immediate follow-up), T3 (4-months post-baseline)
  The DAST is a 10-item brief, self-report instrument for population screening, clinical case finding and treatment evaluation research. It can be used with adults and older youth. The DAST-10 yields a quantitative index of the degree of consequences related to drug abuse. The instrument takes approximately 5 minutes to administer and may be given in either a self-report or interview format. The DAST may be used in a variety of settings to provide a quick index of drug abuse problems. It will be evaluated continuously and as a categorical outcome (yes/no).

SECONDARY OUTCOMES:
Beck Hopelessness Inventory | T1 (baseline, enrollment), T2 (immediate follow-up), T3 (4-months post-baseline)
  This twenty-item measure has been widely used to assess hopelessness through a series of true/false statements (1, 0) that create a sum score.
Anxiety (PROMIS) | T1 (baseline, enrollment), T2 (immediate follow-up), T3 (4-months post-baseline)
  This clinically valid, 7 item measure has been developed as part of the National Institute of Health (NIH) toolkit to assess anxiety in individuals 18 and older. Endpoints range from 1=never to 5=always. It can be used as a sum score and categorizes responses as "none to slight", "mild", "moderate," and "severe".
Depression (PROMIS) | T1 (baseline, enrollment), T2 (immediate follow-up), T3 (4-months post-baseline)
  This clinically valid, 8 item measure has been developed as part of the NIH toolkit to assess depression in the past two weeks. It assesses symptoms ranging from 1=never to 5=always and can be used in individuals 18 and older. It can be used as a sum score and categorizes responses as "none to slight", "mild", "moderate," and "severe".
Loneliness (PROMIS) | T1 (baseline, enrollment), T2 (immediate follow-up), T3 (4-months post-baseline)
  This clinically valid, five item measure was developed as part of the NIH toolkit to assesses feelings of social isolation on a five-point scale from 1=never to 5=not at all.

OTHER OUTCOMES:
Self Compassion Scale | T1 (baseline, enrollment), T2 (immediate follow-up), T3 (4-months post-baseline)
  This twelve-item scale assesses self compassion on a scale of 1=almost never to 5=almost always. Items will be summed and used as a continuous measure.
Difficulties in Emotion Regulation Scale | T1 (baseline, enrollment), T2 (immediate follow-up), T3 (4-months post-baseline)
  This 18-item scale assesses emotion dysregulation on a scale from 1=almost never (0-10%) to 5=almost always (91-100%). It can be summed up (several items reverse coded) and also has six subscales: Nonacceptance of emotional responses, difficulty engaging in goal-directed behavior, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity.
Mindful Attention Awareness Scale | T1 (baseline, enrollment), T2 (immediate follow-up), T3 (4-months post-baseline)
  This is a 15-item scale that assesses mindfulness on a scale of 1=almost always to 6=almost never. It is summed and used as a continuous measure.
Moral Injury and Distress Scale | T1 (baseline, enrollment), T2 (immediate follow-up), T3 (4-months post-baseline)
  This six item scale measures moral injury on a scale from 0=not at all to 4=extremely. It is coded categorically (yes moral injury=1, no moral injury=0) and as a continuous outcome.
Craving | T1 (baseline, enrollment), T2 (immediate follow-up), T3 (4-months post-baseline)
  Craving will be measured for alcohol, opioids, methamphetamine, marijuana, psychedelics or other substances (provide name) from 0=no craving at all to 100=maximum possible.
Trauma-related Shame Inventory | T1 (baseline, enrollment), T2 (immediate follow-up), T3 (4-months post-baseline)
  This 24-item measure assesses trauma-related shame from 0=not true of me to 4=completely true for me. It is summed and analyzed as a continuous outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Prototypes, Pomona, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified, quantitative data will be shared along with a codebook and data dictionary. Data will be completely deidentified.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT06646692/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT06646692/ICF_001.pdf